CLINICAL TRIAL: NCT01982539
Title: An Open-Label Study of the Safety and Efficacy of Zipsor® (Diclofenac Potassium) Liquid Filled Capsules in Pediatric Subjects (Ages 12-17 Years) With Mild to Moderate Acute Pain
Brief Title: Safety and Tolerability of Zipsor® in Pediatric Subjects (Ages 12-17 Years) With Mild to Moderate Acute
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Depomed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 81-0072
Record Dates: First submitted 2013-11-01; First posted 2013-11-13 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Pain
Keywords: pain; NSAID; moderate pain; mild pain; acute pain; mild acute pain; moderate acute pain; mild or moderate acute pain
MeSH Terms: conditions — Pain; Acute Pain; Lymphoma, Follicular | interventions — Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zipsor® (Liquid filled capsules) (Experimental): 25mg/every 6hrs/up to 4 days treatment
  Interventions: Drug: Zipsor®

INTERVENTIONS:
Drug: Zipsor® — Administration of Zipsor® (liquid filled capsules) to patients with mild to moderate acute pain: 25 mg/every 6 hours/up to 4 days treament. Drug taken by mouth.
  Other Names: Diclofenac

SUMMARY:
As part of the PREA(Pediatric Research Equity Act) commitment, the objective of the study is to confirm safety and tolerability of 25 mg of Zipsor® in clinical pediatric subjects.

DETAILED DESCRIPTION:
Open-label study, subjects will be dosed with Zipsor® for the treatment of mild to moderate acute pain for up to 4 days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 12-17 years of age.
* Subjects must be post-op, having mild or moderate acute pain.

Other inclusions apply.

Exclusion Criteria:

* Subject has a known history of allergic reaction, hypersensitivity to diclofenac, aspirin, acetaminophen, or reaction to the non-active ingredients of the study medication.
* Subject has been taking analgesic for 48-72 hours prior to Screening.
* Subject has a history of any GI event greater than 6 months before Screening.
* Subject is currently receiving any medication that is contraindicated for use concomitantly with diclofenac or acetaminophen.
* Subject has previously participated in another clinical study of Zipsor or taking Zipsor for any other indication.
* Subject is requiring treatment for pre-existing hypertension.

Other exclusions apply.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sheffield, Alabama
  - Stanford, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Zipsor® (Liquid Filled Capsules): Administration of Zipsor® (liquid filled capsules) to patients with mild to moderate acute pain: 25 mg/every 6 hours/up to 4 days treatment. Drug taken by mouth.
Period: Overall Study
Arm/Group | Zipsor® (Liquid Filled Capsules)
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Zipsor® (Liquid Filled Capsules)
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.9 (1.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Zipsor® in Pediatric Subjects, Ages 12 to 17 Years
Description: Safety Endpoints:
  * Treatment emergent AEs (TEAEs)
  * Serious adverse events (SAEs)
  * Withdrawals due to AEs
  * Deaths
  * Observed values and changes in vital sign measurements
  * Observed values and changes in clinical laboratory results
  * Physical examination findings
Time Frame: First dose to 30 days after the last dose
Population: The Safety population included all subjects who received at least 1 dose of the study drug.
Measure: Number; unit: participants
Groups:
- Zipsor® (Liquid Filled Capsules): Administration of Zipsor® (liquid filled capsules) to subjects with mild to moderate acute pain: 25 mg/every 6 hours/up to 4 days treatment. Drug taken by mouth.
Arm/Group | Zipsor® (Liquid Filled Capsules)
Number analyzed (Participants) | 25
participants
  Treatment-emergent adverse events (TEAEs) | 12
  Severe TEAEs | 0
  Serious TEAEs | 1
  Serious Adverse Events (SAEs) | 1
  Withdrawals due to AEs | 0
  Deaths | 0

2. Secondary Outcome: Changes in the Numeric Pain Rating Scale (NPRS) Pain Score From Baseline to (1) the First Hour and (2) the Second Hour After the First Dose of Zipsor® Administration.
Description: Numeric Pain Rating Scale (NPRS) measures the subject intensity of pain on an 11-point scale. 0 = No Pain, 10 = Worst Pain at baseline to (1) the first hour and (2) the second hour after the first dose of Zipsor® administration.
Time Frame: From Baseline to 1st and 2nd hour
Population: Full Analysis Set are enrolled patients who had available valid NPRS scores recorded on Day 1, received at least 1 dose of Zipsor, and completed at least 1 postbaseline NPRS score with a valid score. The Full Analysis Set was the primary population for the efficacy analysis. Safety Analysis Set has n=25.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zipsor® (Liquid Filled Capsules)
Number analyzed (Participants) | 23
score on a scale
  Baseline | 4.1 (2.00)
  1st Hour | 2.0 (1.61)
  2nd Hour | 1.7 (1.77)

3. Secondary Outcome: Percentage Difference of Numeric Pain Rating Scale (NPRS) Pain Score From Baseline to (1) the First Hour and (2) the Second Hour After the First Dose of Zipsor® Administration.
Description: as for outcome 2
Time Frame: From Baseline to 1st and 2nd hour
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change of NPRS Score
Arm/Group | Zipsor® (Liquid Filled Capsules)
Number analyzed (Participants) | 23
Percent Change of NPRS Score
  Percent Change from baseline to 1 hour postdose | -55.32 (24.899)
  Percent Change from Baseline to 2 hours post dose | -60.25 (41.549)

ADVERSE EVENTS:
Arm/Group | Zipsor® (Liquid Filled Capsules)
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 9/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zipsor® (Liquid Filled Capsules) (N=25)
Post Procedural Bile Leak (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zipsor® (Liquid Filled Capsules) (N=25)
Nausea (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees that sponsor shall have the right to the first publication of the study results which is intended to be a joint, multi-center publication. Following the first publication, the PI may publish study data or results, provided however PI submits the proposed publication to sponsor for review at least 60 days prior to the date of the proposed publication. Sponsor may remove any information that is considered confidential and / or proprietary other than study data.